CLINICAL TRIAL: NCT05784324
Title: COMPRESSED - A Longitudinal Study of Compressed Work Schedules Within the Health, Care and Welfare Services
Status: Not yet recruiting | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Collaborators: The Research Council of Norway (Other); University of Oslo (Other); Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: 202316
Record Dates: First submitted 2022-12-20; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-12

CONDITIONS: The Focus of the Study is Shift Work

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Employees within the municipal health, care and welfare services: All employees within the municipal health, care and welfare services. No internvention. We investigate the relationship between caracteristics of their shift systems and potential outcomes.
  Interventions: Other: No intervention
- Employees within the municipal health, care and welfare services 2: Employees within the municipal health, care and welfare services, replying to a survey. Sample is drawn by representative unions. No internvention. We investigate the relationship between caracteristics of their shift systems and potential outcomes.
  Interventions: Other: No intervention
- Users of the municipal health, care and welfare services.: Users of the municipal health, care and welfare services.No internvention. We investigate the relationship between caracteristics of the shift systems worked and potential outcomes for users.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of COMPRESSED is to investigate the potential consequences of a compressed work schedule within the municipal health, care and welfare services.

DETAILED DESCRIPTION:
The aim of COMPRESSED is to investigate the potential consequences of a compressed work schedule within the municipal health, care and welfare services.

A compressed work schedule is defined by an increase in numbers of hours per day, and a reduction of number of days per week. Compressed work schedules are advocated as a tool to reduce involuntary part-time contracts, and improve employee recruitment and retention, as well as improve employee health and quality of care.

However, the empirical support of such claims is limited, mixed, and suffers from several methodological shortcomings. There is a clear lack in studies investigating the potential moderating and mediating mechanisms, despite moderating variables such as shift intensity being likely to have an impact. In collaboration with unions and employers, COMPRESSED uses a longitudinal mixed method design, to investigate the short- and long-term consequences of compressed work schedules, as well as potential moderating and mediating variables. Each of the research questions will be addressed with complimentary methods in each of the work packages.

The project COMPRESSED will examine:

In-depth narrative interviews eliciting employees', employers', and patients'/users' own perceptions of consequences, moderators and mechanisms.

A retrospective intervention study using registry data, examining compressed work schedules implemented over the past 5 years.

A two year longitudinal survey looking at long-term effects and 4) a diary study across two weeks, looking at short-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Employed within the municipal health, care and welfare services.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Employes within the municipal health, care and welfare service
Sampling Method: Non-Probability Sample
Enrollment: 700000 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Featigue | 2027
  Fatigue General Fatigue scale from the Checklist of Individual Strength (CIS-20; Vercoulen et al., 1994)
Mental health | 2027
  Hopkins Symptom Checklist (SCL-5)
Generell helse | 2027
  The general health measure from the Short-Form Health Survey (SF-36) (Ware, 1992)
Sickness absence | 2027
  self-repport and regestry data
Quality of care | 2027
  From COPSOQ
Care left undone | 2027
  adapted from (Senek et al., 2020) and a measure by (Ball, Murrells, Rafferty, Morrow, & Griffiths, 2014) informed by the validated Basel Extent of Rationing of Nursing scale (Schubert et al., 2008).
Intention to quit | 2027
  (Kuvaas, 2006).
Occupational commitment | 2027
  (Tam, Korczynski, & Frenkel, 2002)
Regestry-data | 2027
  We will attempt to measure 1. Health, 2 recruitment and retention and 3. Quality of care, using registry data. And important part of the project will be to explore how these aspects are best measured using registry data. Their final operationalization is therefore not set.

IPD SHARING:
Plan to Share IPD: No